CLINICAL TRIAL: NCT00170703
Title: Assessment of the Safety and Effectiveness of Targeted Sub-Threshold Epidural Cortical Stimulation Delivered Concurrent With Speech-Language Rehabilitation to Enhance Recovery in Patients Suffering From Broca's Aphasia, Following a Stroke.
Brief Title: Assessment of Cortical Stimulation Combined With Rehabilitation to Enhance Recovery in Broca's Aphasia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northstar Neuroscience (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V0325
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Stroke; Broca's Aphasia
Keywords: Cortical Electrical Stimulation; Ischemic Stroke; Broca's Aphasia; Speech Rehabilitation; Functional MRI
MeSH Terms: conditions — Stroke; Aphasia, Broca; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cortical Electrical Stimulation

SUMMARY:
The primary objective of this feasibility study is to evaluate the safety and effectiveness of targeted sub-threshold epidural cortical stimulation delivered concurrent with speech-language rehabilitation activities to enhance recovery in study subjects suffering from Broca's aphasia (the inability to speak or to organize the muscular movements for speech), following a stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the most common cause of disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. Approximately 150,000 to 250,000 stroke survivors becoming severely and permanently disabled each year.

A common neurological deficit among these stroke survivors, and thus a substantial contributor to post-stroke disability is Broca's aphasia, a condition in which the patient is unable to speak normally, as they cannot effectively organize the muscular movements required for speech. Broca's aphasia is often referred to as "non-fluent" or "motor" aphasia as essentially the patient has impaired motor abilities for speech and thus, become non-fluent in speech/language. The loss of speech for these patients is extremely debilitating and has enormous social and economic impact to the quality of life for these patients. Presently, the only treatment available for patients with Broca's aphasia is speech-language rehabilitation. However, with rehabilitation only, many patients achieve a less than satisfactory improvement in speech-language function and thus, are left with significant disability.

Since Broca's aphasia is largely due to an impairment of language-related motor function, researchers and clinicians believe it is very likely that cortical stimulation in conjunction with speech rehabilitation may also enhance recovery of language motor function for Broca's aphasia patients. This study proposes to evaluate the safety and effectiveness of such cortical electrical stimulation in study subjects with Broca's aphasia after stroke, delivered concurrent with speech-language rehabilitation.

In addition to evaluating changes from baseline level, safety and efficacy measures will be compared to patients who undergo the same speech-language rehabilitation activities but without cortical stimulation. The two study groups will be compared to determine the degree to which the aphasia can be improved beyond rehabilitation alone by epidural stimulation of a targeted cortical region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an ischemic stroke.
* Subjects must have a language dominant left hemisphere.
* Subjects must be diagnosed as having predominantly Broca's aphasia.
* Age 21 years or older.

Exclusion Criteria:

* Primary hemorrhagic stroke.
* Any additional stroke associated with incomplete speech recovery.
* Any neurologic or physical condition that impairs speech function.
* History of seizure disorder.
* Global aphasia or inability to participate in routine speech therapy.
* Untreated or inadequately treated depression.
* History of traumatic brain injury, or spontaneous subdural or epidural hematoma that has resulted in a fixed (stable) speech-language deficit.
* Major active psychiatric illness that may interfere with required study procedures.
* Contraindication to magnetic resonance (MR) imaging.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2004-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Aphasia Quotient on the Western Aphasia Battery (WAB-AQ) at follow-up week 1
Measures of speech rate obtained from Language Sample Analysis at follow-up week 1

SECONDARY OUTCOMES:
Serious Adverse Event rate at follow-up weeks 1, 6 & 12-week
Aphasia Quotient on the Western Aphasia Battery (WAB-AQ) at follow-up weeks 6 & 12
Measures of speech rate obtained from Language Sample Analysis at follow-up weeks 6 & 12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Univ. of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Cherney LR. Epidural Cortical Stimulation as Adjunctive Treatment for Nonfluent Aphasia: Phase 1 Clinical Trial Follow-up Findings. Neurorehabil Neural Repair. 2016 Feb;30(2):131-42. doi: 10.1177/1545968315622574. Epub 2015 Dec 23. PMID 26704258